CLINICAL TRIAL: NCT02867553
Title: Multiple Fields Radiotherapy Versus Intravenous Rituximab in the Treatment of Indolent Cutaneous Lymphomas B-cell With Multiple or Recurrent Lesions
Acronym: RADIO-LYMPH
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PN09001
Record Dates: First submitted 2016-08-11; First posted 2016-08-16 (Estimated); Last update posted 2016-09-07 (Estimated); Status verified 2016-09

CONDITIONS: Indolent Cutaneous B Cell Lymphomas
MeSH Terms: interventions — Rituximab

ARMS (2):
- Rituximab by intravenous (Experimental): attack treatment (4 slow intravenous perfusions of rituximab at a dose of 375 mg / m2 on day 1, day 8, day 15 and day 22) and maintenance treatment (intravenous perfusions of rituximab at a dose of 375 mg / m2 every 2 months for 2 years).
  Interventions: Drug: rituximab
- multi-field radiotherapy (Active Comparator): multi-fields radiotherapy with a dose between 20 and 30 gray and a fractionated dose over 2 at 3 weeks.
  Interventions: Radiation: Multi-fields radiotherapy

INTERVENTIONS:
Drug: rituximab
  Arms: Rituximab by intravenous
Radiation: Multi-fields radiotherapy
  Arms: multi-field radiotherapy

SUMMARY:
Cutaneous lymphomas are the most frequent extranodal lymphomas after digestive lymphomas. A quarter are B-cell lymphomas. 80% of cutaneous B cell lymphomas are indolent cutaneous B cell lymphomas. These indolent cutaneous B cell lymphomas are characterized by good prognosis (survival rate at 5 years: 90%), but also by the frequency of cutaneous recurrences. The radiotherapy is currently the most widely used treatment, with complete response rate close to 100% for a lesion treated. However, it has limits when there are outset multiple lesions inaccessible to a single radiotherapy field (concerning one case in three), or during recurrences. In these situations, conventional chemotherapy is not recommended and multi-field radiotherapy is often used empirically, but its effectiveness has never been studied prospectively.

Recently, retrospective studies with small numbers patients (totaling sixty patients) reported complete response rates of 80 to 100% with rituximab (anti-cluster of differentiation antigen 20 (CD20) antibodies) used as monotherapy in non-standardized treatment by intravenous with a recurrence rate of less than one case in three. These data suggest that rituximab by intravenous with a standardized initial cycle followed by a maintenance therapy could improve the prognosis of indolent cutaneous B cell lymphomas with multiple lesions or of recurrent lesions.

DETAILED DESCRIPTION:
Compare the efficacy and safety of two treatment strategies for indolent cutaneous B cell lymphomas with multiple or recurrent lesions: Rituximab by intravenous versus multi-field radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* patients with histological diagnosis of indolent cutaneous B cell lymphomas
* patients with multiple lesions inaccessible to a single field of radiotherapy or patients with a recurrence outside the field of first radiotherapy
* patient with a lesion of at least 15 mm in major axis and a total tumor surface area greater or egal than 4 cm2
* patient with a negative staging
* patient consenting to participate to the study
* patient enrolled in the national healthcare insurance program
* patient older than 18 years

Exclusion Criteria:

* contraindication for rituximab or radiotherapy
* immunosuppressive therapy
* immunosuppression

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2011-10; Primary Completion 2018-07 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Disease free survival | 5 years
  Disease free survival

CONTACTS AND LOCATIONS:
Locations (1):
- Chu de Reims, Reims, France, France